CLINICAL TRIAL: NCT00812370
Title: An Open-label, Dose-finding, Pharmacokinetic, Safety and Efficacy Study of Bivalirudin in Children Between 6 Months and 18 Years of Age
Brief Title: The UNBLOCK Study: Utilization of Bivalirudin On Clots in Kids
Acronym: UNBLOCK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Baylor College of Medicine (Other); Children's Hospital Colorado (Other); Children's Hospital of Philadelphia (Other); Nationwide Children's Hospital (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Guy Young, Director, Hemostasis and Thrombosis Center, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3070850
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Deep Venous Thrombosis
Keywords: DVT; Deep Venous Thrombosis; UNBLOCK; Bivalirudin; Angiomax
MeSH Terms: conditions — Venous Thrombosis | interventions — bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label (Experimental)
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — The initial bolus dose will be 0.125 mg/kg followed immediately by a continuous infusion of 0.125 mg/kg/hour.
  Other Names: Angiomax

SUMMARY:
Thrombosis is a significant medical complication in children with chronic diseases. The currently utilized treatments have many drawbacks which can lead to poor outcomes. More modern therapies are available but have not been systematically tested in children. This study will determine whether one such medication, bivalirudin is a safer and more effective alterative.

This study will monitor what effects the drug has upon the child's body and how the body processes the study drug (absorption, metabolism and elimination). The study will also evaluate the drug's effectiveness by following how long it takes to dissolve the clot. The safety issues being monitored relate to any observations of major or minor bleeding episodes after taking the drug, and/or any other side effects.

DETAILED DESCRIPTION:
This will be an open-label, single-arm, dose-finding, pharmacokinetic, safety and efficacy study of bivalirudin in children 6 months to 18 years of age with deep vein thrombosis. The specific aims are as follows:

1. Pharmacodynamic analysis based on the activated partial thromboplastin time (aPTT) will be performed and the best bolus dose and initial infusion dose of bivalirudin will be determined for 3 age cohorts of children.
2. Pharmacokinetic analysis of bivalirudin will be determined based on bivalirudin plasma levels in the same 3 age cohorts.
3. Comparison of pharmacokinetics with pharmacodynamics will be performed to determine whether the aPTT is an adequate surrogate for plasma bivalirudin levels.
4. The rate of clot resolution within 48-72 hours will be determined.
5. The safety of bivalirudin will be determined by assessing for major and minor bleeding and other adverse events.

A total of 30 patients will be enrolled in this study. They will be divided into 3 groups according to their age range (6 months-age to > 5, 5 to > 12 years and 12 to >18 years). The patient must have a deep vein thrombosis (clot in an artery or vein) that has been seen on an imaging test. After receiving the study drug, the subjects will then have blood tests at specific timepoints to measure how the drug is effecting the body and how the drug is acting once it is in the body. Based upon the levels of the blood tests, the dose of the study drug may be adjusted or stopped. The subject will continue on the drug until the clot is dissolved, the subject is prescribed a different anticoagulant or the physician or parents decide to remove the child off of the study. The drug will also be discontinued if any excessive bleeding or severe side effects related to the drug are observed. A follow up imaging study will be performed on all patients 48-72 hours after the drug was started. If the clot is still present at this time, another imaging study will be done at 30 days after the drug was given. The subjects will continue to have lab tests twice weekly for about 3 weeks to monitor for the effects of the drug. After completion of the study, the patient will undergo a study exit physical exam between 20-40 days after the drug was stopped.

ELIGIBILITY:
Inclusion Criteria:

* Children > 6 months to < 18 years of age.
* Deep vein thrombosis demonstrated by objective testing (Duplex ultrasonography, venography, CT venography, MR venography, echocardiography). This imaging must be performed within 72 hours prior to initiation of study drug if no other anticoagulation has been started. If receiving other anticoagulation prior to start of study drug, imaging must be performed within 24 hours of study drug initiation.
* Informed consent and assent from parent/guardian/patient

Exclusion Criteria:

* Treatment of present thrombus with thrombolytic agent.
* Treatment of present thrombus with another anticoagulant for more than 48 hours (low dose heparin for maintenance of venous or arterial catheter patency is allowed).
* Baseline prothrombin time (PT) which is more than 3 seconds above the upper limit of normal or baseline activated partial thromboplastin time (aPTT) which is more than 5 seconds above the upper limit of normal.
* Creatinine which is more than 20% above the upper limit of normal for age.
* Presence of a known bleeding disorder.
* Active bleeding.
* Planned invasive procedure within 3 days.
* Known pregnancy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The study will assess efficacy by re-evaluating thrombus at 48-72 hours as well as continued efficacy by re-evaluating the thrombus at ~30 days after study drug initiation. | 30 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) will also be assessed by measuring plasma bivalirudin levels and correlation of the PD to the PK parameter will be performed. The study will also assess safety by evaluating for bleeding, as well as other adverse events. | twice a week until drug discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Guy A Young, MD, Principal Investigator — CHLA
Locations (6):
- United States (6):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCD Hemophilia & Thrombosis Center, Aurora, Colorado
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Childrens Hospital of Philidelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas